CLINICAL TRIAL: NCT01002222
Title: Open-Label, Six-Month Extension of Protocol MCS-2-TWN-a to Further Evaluate the Efficacy and Safety of MCS-2 for the Treatment of Lower Urinary Tract Symptoms Suggestive of Benign Prostatic Hyperplasia in Treatment Naïve Male Subjects
Brief Title: Open-Label Extension Study of MCS-2 in the Treatment of Lower Urinary Tract Symptoms (MCS-2-US-c)
Acronym: MCS-2-US-c
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Health Ever Bio-Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCS-2-US-c
Record Dates: First submitted 2009-10-25; First posted 2009-10-27 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Lower Urinary Tract Symptoms; Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; MCS-2; Multi-Carotenoids; Lower Urinary Tract Symptoms; International prostate symptom score
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MCS-2 (Experimental)
  Interventions: Drug: MCS-2

INTERVENTIONS:
Drug: MCS-2 — 15 or 30 mg/day of MCS-2 soft-gel capsules Qd for 24 weeks, depending on which dose level is selected after the phase 2b part of the protocol MCS-2-US-a.
  Other Names: MUS

SUMMARY:
This is an open-label extension study of another study protocol, MCS-2-US-a. Subjects who have completed the 12-week treatment and procedures under the protocol MCS-2-US-a will be eligible for this study.

DETAILED DESCRIPTION:
This open-label extension study is designed to further assess the long-term safety and efficacy of MCS-2. Subjects who have completed the 12-week treatment and procedures under the protocol MCS-2-TWN-a will be eligible for another 40 weeks of MCS-2 treatment at the optimal dose selected after the phase 2b part of MCS-2-US-a. Subjects are limited to those who are currently not being treated medically for BPH or LUTS.

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed 12 weeks of treatment under the protocol MCS-2-US-a.
* Subject is able to understand and willing to conform to the study procedures and has signed the informed consent form for participation in this extension study.

Exclusion Criteria:

* Subject has severe LUTS at the last visit under the protocol MCS-2-US-a.
* Subject is considered ineligible for the study by the investigator(s).

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAE) | 36 weeks

SECONDARY OUTCOMES:
Changes from baseline in International Prostate Symptom Score (I-PSS) | 36 weeks
Changes from baseline in urine flow rate | 36 weeks
Changes from baseline in serum lycopene levels | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Allan J Pantuck, MD, MS, FACS, Principal Investigator — University of California, Los Angeles
Locations (1):
- David Geffen School of Medicine at UCLA, Los Angeles, California, United States